CLINICAL TRIAL: NCT06709378
Title: Effectiveness and Safety of 25-Gauge Needle-Assisted Phacoemulsification of Dislocated Intravitreal Lens Nucleus
Status: Completed | Type: Observational
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Qing Feng, Principal Investigator, Changzhou No.2 People's Hospital
Other Study IDs: 213000
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Dislocated Lens; Pars Plana Vitrectomy; Phacoemulsification; Needle
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The goal of this observational study is to learn about the effects of 25-gauge (G) needle-assisted phacoemulsification to remove dislocated intravitreal lens nuclei.

DETAILED DESCRIPTION:
Patients with dislocated intravitreal lens nuclei who underwent 23G pars plana vitrectomy (PPV) and 25G needle-assisted phacoemulsification between July 2022 and September 2024 were included. Primary outcomes included best-corrected visual acuity (BCVA) and intraocular pressure (IOP). Secondary outcomes included corneal endothelial cell count (CECC) and the incidence of intraoperative and postoperative complications. These outcomes were statistically analyzed both preoperatively and postoperatively. A minimum follow-up of 6 months was completed for all eyes.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of dislocated intravitreal lens nuclei Signed informed consent

Exclusion Criteria:

Surgical contraindications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dislocated intravitreal lens nuclei who underwent 23G pars plana vitrectomy (PPV) and 25G needle-assisted phacoemulsification and without surgical contraindications exist.
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | Preoperatively and postoperatively for at least 6 months.
  Best corrected visual acuity was measured with logarithmic visual acuity chart.

SECONDARY OUTCOMES:
Intraocular pressure | Preoperatively and postoperatively for at least 6 months.
  Intraocular pressure was measured with noncontact tonometer.
Corneal endothelial cell count | Preoperatively and postoperatively for at least 6 months.
  Corneal endothelial cell count was measured with specular microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Xincheng Sun, Study Director — Changzhou No.2 People's Hospital
Locations (1):
- the Second People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No